CLINICAL TRIAL: NCT06475040
Title: Accelerated Intermittent Theta Burst Stimulation to a Novel DLPFC Target for Anxiety and Trauma-related Disorders: a Pilot Study
Brief Title: TMS for Anxiety and Trauma-related Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRCui
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-05

CONDITIONS: Anxiety Symptoms; Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open-label aiTBS to novel right dmPFC TMS anxiety target (Experimental)
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — non-invasive form of brain stimulation accelerated intermittent theta burst stimulation (aiTBS)

SUMMARY:
The present pilot study will apply accelerated intermittent theta burst stimulation (aiTBS) to a novel transcranial magnetic stimulation (TMS) target for anxiety derived via causal network mapping.

DETAILED DESCRIPTION:
Anxiety-related disorders represent the most common class of mental-health disorders and are associated with high rates of non-response and relapse to current treatments. Transcranial magnetic stimulation (TMS) applied to the dorsolateral prefrontal cortex (dlPFC) has been shown to reduce anxiety comorbid with major depressive disorder (MDD). However, anxiety-specific targets have received insufficient attention.

An anxiety specific transcranial magnetic stimulation (TMS) target was recently derived via causal network mapping and was shown to reduce anxiety versus depression symptoms to a greater extent than the conventional dlPFC target in an MDD sample with comorbid anxiety. While potentially promising, this target has yet to be trialed in an anxiety-related disorder sample.

The current open-label study will be the first to evaluate the preliminary effectiveness and safety of this novel right dorsomedial prefrontal cortex (dmPFC) TMS target. MRI-guided neuronavigation will be used to locate this target in each participant. An accelerated intermittent theta-burst (aiTBS) dosing regimen will be used. Based on a 90% resting motor threshold (adjusted for cortical depth), 50 sessions of iTBS will be administered (1800 pulses per session, with a 50-minute inter-session interval) and delivered in a schedule of 10 sessions per day for 5 consecutive days. Clinical assessments and resting-state functional MRI scans will be conducted before and after aiTBS. Heart rate variability (HRV) and eye-movement measures will be collected before and after aiTBS.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of generalized anxiety disorder (GAD), social anxiety disorder (SAD), panic disorder (PD), and/or post-traumatic stress disorder (PTSD) as defined by DSM-5 criteria.
2. Male or female between 18 and 60 years old.
3. Right-handed.
4. Can understand and sign an informed consent document.
5. Beck Anxiety Inventory (BAI) score of 16 or higher.
6. On a stable medication/psychotherapy regimen for at least 6 weeks prior to baseline visit and throughout the duration of the study.
7. In good general health, as ascertained by medical history.
8. Pharmacological treatment resistance or psychotherapeutic treatment resistance.

Exclusion Criteria:

1. Substance use disorders, eating disorders, significant suicidal ideation, mental disorder due to a medical or neurocognitive condition, lifetime psychosis, bipolar disorder, developmental disorders.
2. History of brain surgery and epilepsy.
3. Presence of metallic foreign bodies, such as cardiac pacemakers and stents.
4. Any medical condition or medication that increases the risk of seizures.
5. Pregnancy.
6. Intellectual disability.
7. Current severe somatic disease, such as cancer, heart failure, pneumonia, etc.
8. Severe claustrophobia that prevents the use of MRI.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Effectiveness as measured by Beck Anxiety Inventory | Anxiety symptoms will be measured before the TMS treatment, immediately after 5 days of TMS, 1 week and 4 weeks respectively after completion of the TMS treatment
  Measure of severity of anxiety - total score of Beck Anxiety Inventory ranges from 0 to 63 (higher numbers indicate higher severity)

SECONDARY OUTCOMES:
Safety as measured by number of participants with Adverse Events | Each afternoon after treatment during the 5 days of treatment
  Count of Adverse Events Reported during follow up
Resting-state functional MRI (rsfMRI) scan | Baseline (before treatment) and after 5 days of TMS stimulation
  Functional MRI scan will be conducted before and after treatment to assess for treatment-induced changes in brain connectivity
Hamilton Anxiety Rating Scale (HAMA) | Baseline (before treatment), 5 days of TMS treatment, and 1 and 4 weeks after the end of the TMS stimulation
  Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56
State-Trait Anxiety Inventory (STAI) | Baseline (before treatment), 5 days of TMS treatment, and 1 and 4 weeks after the end of the TMS stimulation
  State and trait anxiety will be assessed separately with 20 respective questions. Scores range from 20 to 80, with higher scores indicating greater anxiety
Hamilton Depression Rating Scale (HAMD) | Baseline (before treatment), 5 days of TMS treatment, and 1 and 4 weeks after the end of the TMS stimulation
  Measure of depression severity - total score of Hamilton Depression Scale ranges from 0 (no depression) to 60 (most severe depression)
Sheehan Disability Scale (SDS) | Baseline (before treatment), 5 days of TMS treatment, and 1 and 4 weeks after the end of the TMS stimulation
  Three domains can be summarized to evaluate global functional impairment by adding the scores of each, resulting in global SDS score ranges from 0 (unimpaired) to 30 (highly impaired)

CONTACTS AND LOCATIONS:
Overall Officials: Huiru Cui, Ph.D, Principal Investigator — Shanghai Mental Health Center, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No